CLINICAL TRIAL: NCT03752307
Title: Double-blind, Placebo-controlled, Randomized Study of the Safety and Tolerability of Isoxsuprine HCL Combined With High Dose Steroid Treatment of Multiple Sclerosis (MS) Relapse
Brief Title: Safety and Tolerability of ISX (Isoxsuprine HCL) in MS Relapses
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of New Mexico (Other)
Responsible Party: Principal Investigator, Corey C Ford, MD, PhD, Senior Associate Dean for Research, Office of Research, University of New Mexico
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18-643
Record Dates: First submitted 2018-11-15; First posted 2018-11-23 (Actual); Results first posted 2024-02-06 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-01

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Isoxsuprine; Adrenal Cortex Hormones; Methylprednisolone; Prednisone

STUDY DESIGN:
Intervention Model Description: This is a proof of concept, randomized, double-blind, placebo-controlled, 2-arm, parallel group study of Isoxsuprine in MS subjects experiencing a typical relapse
Who Masked: Participant, Investigator
Masking Description: Subjects will be randomized 1:1 according to a computer-generated allocation scheme to receive either Isoxsuprine HCL 1 capsule 3 times daily for 5 days or matching placebo.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Corticosteroid & Isoxsuprine HCL (Experimental): Corticosteroid pulse of either daily iv methylprednisolone 1000 mg/day or 600mg oral prednisone two times a day at approximately 8AM and noon for 3 to 5 consecutive days and Isoxsuprine Hydrochloride one 10 mg Capsule 3 times daily for 5 consecutive days
  Interventions: Drug: Isoxsuprine Hydrochloride; Drug: Corticosteroid
- Corticosteroid & Placebo (Placebo Comparator): Corticosteroid pulse of either daily iv methylprednisolone 1000 mg/day or 600mg oral prednisone two times a day at approximately 8AM and noon for 3 to 5 consecutive day and placebo one Capsule 3 times daily for 5 consecutive days
  Interventions: Drug: Placebo; Drug: Corticosteroid

INTERVENTIONS:
Drug: Isoxsuprine Hydrochloride — Compounded Isoxsuprine hydrochloride capsules
  Other Names: Duvadilan
  Arms: Corticosteroid & Isoxsuprine HCL
Drug: Placebo — Identical microcrystalline cellulose placebo manufactured to mimic Isoxsuprine Hydrochloride 10 MG capsules
  Arms: Corticosteroid & Placebo
Drug: Corticosteroid — This can be any accepted regimen, including daily iv methylprednisolone 1000 mg/day or 600mg oral prednisone two times a day at approximately 8AM and noon
  Other Names: Methylprednisolone; Prednisone

SUMMARY:
This is a proof of concept, randomized, double-blind, placebo-controlled, 2-arm, parallel group study of Isoxsuprine in MS subjects experiencing a typical relapse.

Evidence from preclinical stroke models and experimental allergic encephalomyelitis suggest that isoxsuprine hydrochloride may have neuroprotective activity and reduce disability in animal models. Given its potential neuroprotective effects in CNS injury models, the investigators propose to test it as a safe, tolerable add on treatment for acute relapses in patients with relapsing forms of MS.

DETAILED DESCRIPTION:
This is a proof of concept, randomized, double-blind, placebo-controlled, 2-arm, parallel group study of Isoxsuprine in MS subjects experiencing a typical relapse.

All subjects will have a documented diagnosis of relapsing MS or a clinically isolated syndrome by international criteria. The relapse will be of sufficient severity that their physician recommends treatment with a high dose corticosteroid pulse. All subjects will have a physical examination and history with questions on drug sensitivities. Subjects experiencing the onset of objective neurological deficits consistent with relapse within 7 days of randomization are eligible for screening for this study. Those currently on MS disease modifying therapy will have received a stable regimen of the medications for at least 30 days prior to screening and will continue the same doses and regimens for the duration of their study participation.

Consented subjects will be assessed for relapse criteria and those who meet study eligibility criteria and agree to be treated with a standard 3 to 5 day pulse of high dose corticosteroids, will be randomized with equal probability to 1 of 2 treatment groups: placebo capsule or active Isoxsuprine (ISX).

The Screening Visit will take place within 7 days of relapse onset and within 48 hours of initiating high dose steroids. Subjects may start corticosteroids anytime during this 7 day window. During the screening period, subjects will be assessed with the Expanded Disability Status Scale (EDSS), Multiple Sclerosis Functional Composite (MSFC), and cognitive testing prior to treatment with ISX or placebo (1:1 ratio). Safety Assessments during screening will include a physical exam, electrocardiogram, vital signs, weight and a urine pregnancy test for females of child bearing potential. At 7 (± 1) days following the completion of the 5-day ISX dosing, subjects will be re-assessed with the EDSS.

Subjects will be evaluated for treatment response using the EDSS and other standard measures.

Study drug will be administered as one (1) 10 mg capsule, 3 times daily for 5 days in conjunction with concomitant dosing with high dose corticosteroids. This can be any accepted regimen, including daily iv methylprednisolone 1000 mg/day or 600mg oral prednisone two times a day at approximately 8AM and noon, with food, as typically provided by UNM MS Specialty Clinic.

ELIGIBILITY:
Inclusion Criteria:

* 1. Subjects must be adequately informed and understand the nature and risks of the study and must be able to provide a signature and date on the ICF; 2. Male or female subjects between 18 and 50 years of age, inclusive; 3. Confirmed diagnosis of Multiple Sclerosis or Clinically Isolated Syndrome (CIS) suggestive of MS, according to the 2010 Revised McDonald criteria.

  4. On a stable regimen of medications taken specifically to treat MS for at least 30 days prior to screening, and willing to continue the same doses and regimens for the duration of study participation; 5. New neurological disability consistent with MS relapse no longer than 7 days prior to screening; 6. Screen visit and randomization must occur within 48 hours of subject initiating steroid treatment.

  7. Maximum EDSS score during screening of 6.5; 8. Sufficient ambulatory ability (ambulatory aids acceptable if used consistently) to complete two trials of the Timed 25 Foot Walk (T25FW) at the screening visit with the two trials completed within 5 minutes of each other in accordance with the specific instructions provided by the National MS Society Functional Composite Manual.

  9. Subject must be willing to take a high dose steroid (600mg oral prednisone two times a day (bid).

  10. Subjects must have a mean systolic blood pressure ≤ 160 and greater than 100 mm Hg and a mean diastolic blood pressure of ≤ 100 and greater than 50 mm Hg determined by the average of 3 seated readings taken at least 5 minutes apart at the Screening Visit.

  11. Subjects must be able to communicate effectively with study personnel. For this reason only English speaking subjects will be eligible for the study.

  12. Subjects must be able and willing to follow all protocol requirements and study restrictions.

  13. Subjects must be able and willing to return for all study visits.

Exclusion Criteria:

* 1. Subject is from a vulnerable population, as defined by the US CFR Title 45, Part 46, Section 46.111(b) and other local and national regulations, including but not limited to, employees (temporary, part-time, full time, etc) or a family member of the research staff conducting the study, or of the sponsor, or of the IRB.

  2. Subject has only sensory, bowel/bladder, and/or cognitive symptoms of MS associated with the most recent relapse.

  3. Subject has cognitive or behavioral impairment that in the opinion of the investigator would impair the ability of the subject to comply with study procedures.

  4. Subject has any known contraindication(s) to the use of corticosteroids or isoxsuprine hydrochloride (ISX), including, but not limited to:
  * any current uncontrolled hypertension, primary adrenocortical insufficiency
  * Any current psychoses, infectious disease, or Cushing's syndrome.
  * Any current congestive heart failure (defined as New York Heart Association (Functional Class III to IV).
  * Peptic ulcer (within 24 weeks prior to the Screening Visit).
  * Recent major surgery (within 24 weeks prior to the Screening Visit).
  * Use of tizanidine any time in the past 30 days. 5. Subject has a clinically significant infection requiring intravenous administration of antibiotics and hospitalization prior to the Screening Visit.

    6. Subject has poorly controlled type 1 or type 2 diabetes mellitus (prior diagnosis of gestational diabetes mellitus is not exclusionary 7. Received systemic steroids for a problem unrelated to the MS relapse within 30 days prior to screening.

    8. History of other neurological disease that, 'in the opinion of the Investigator, would affect motor function or cognition; 9. For patients with a history of Major Depressive Disorder, at risk for worsening depression due to steroids or the presence of active depressive symptoms sufficient, in the opinion of the investigator, to affect the subject's ability to complete study assessments, or which would not be in the subject's best Interest to participate in the study; 10. Presence of cognitive impairment sufficient, in the opinion of the investigator, to affect the subject's ability to complete study assessments, or which would not be In the subject's best interest to participate in the study 11. History of sensory impairments (e.g., hearing, vision) that, In the opinion of the investigator, would impair the subject's ability to complete study assessments; 12. History of current alcohol or substance abuse or dependence; 13. History of myocardial infarction, or NYHA Functional Classification of Heart Failure Class 3 or 4 within 2 years prior to screening, or history of coronary artery disease and/or active angina pectoris; 14. Any clinically significant ECG abnormalities;; 15. Inability to swallow oral capsules, or a history of gastrointestinal malabsorption that would preclude the use of oral medication; 16. If female, is pregnant or lactating; 17. History of hypersensitivity or allergic reaction to any of the study drugs. 18. History of heavy use of tobacco/smoking

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2019-02-15 (Actual); Primary Completion 2023-07-06 (Actual); Study Completion 2023-07-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Corey C Ford, M.D., Ph.D., Principal Investigator — University of New Mexico
Locations (1):
- University of New Mexico MS Specialty Clinic, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Corticosteroid & Isoxsuprine HCL | Corticosteroid & Placebo
Started | 1 | 1
Completed | 1 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Corticosteroid & Isoxsuprine HCL | Corticosteroid & Placebo | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] — Data collected was only from 1 participant and therefore no data range available to report.
  years | 25 [25 to 25] | 26 [26 to 26] | 25.5 [25 to 26]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 0 | 1
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Treatment-Emergent Adverse Events in Subjects by Measuring Measuring Changes in Vital Signs
Description: Vital Signs: Blood pressure greater than 140/90, pulse greater than 110 and temperature greater than 37.8 Celsius.
Time Frame: Baseline to Week 12
Measure: Number; unit: Adverse Events
Arm/Group | Corticosteroid & Isoxsuprine HCL | Corticosteroid & Placebo
Number analyzed (Participants) | 1 | 1
Adverse Events | 0 | 0

2. Secondary Outcome: Incidence of Adverse Event Expanded Disability Status Scale (EDSS)
Description: The unit of measure is 0 (no disability) to 10 (death). An increase in EDSS score from baseline measure during with steroid/study treatment during the study would be considered an adverse event.
Time Frame: Baseline to Week 12
Measure: Number; unit: Adverse Events
Arm/Group | Corticosteroid & Isoxsuprine HCL | Corticosteroid & Placebo
Number analyzed (Participants) | 1 | 1
Adverse Events | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the 12 week study duration. Any serious adverse events that occurred were followed until they had resolved or stabilized.
Description: Adverse events were not related to the study drug and did not occur in an unanticipated manner.
Arm/Group | Corticosteroid & Isoxsuprine HCL | Corticosteroid & Placebo
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 1/1 | 0/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Corticosteroid & Isoxsuprine HCL (N=1) | Corticosteroid & Placebo (N=1)
Heart burn and Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-06-18): https://cdn.clinicaltrials.gov/large-docs/07/NCT03752307/Prot_000.pdf
  • Informed Consent Form (2020-06-18): https://cdn.clinicaltrials.gov/large-docs/07/NCT03752307/ICF_001.pdf